CLINICAL TRIAL: NCT04704765
Title: The Effectiveness of Abdominal Breathing Training on Reducing Anxiety
Brief Title: Abdominal Breathing Training on Reducing Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Xuan-Yi Huang, RN, DNSc, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200105R
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anxiety
Keywords: Abdominal Breathing Training, Anxiety, Effectiveness
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Using an experimental randomized controlled trial approach. The experimental group receiving abdominal breathing training, and control group without training. The effectiveness assessment used the Beck anxiety inventory, required to be completed by both the experimental group and control group. This study performed the pre-and-post assessments. This study performed the pre-test before the implementation of abdominal breathing training, and performed the post-test at Week 4 and Week 8 the end of abdominal breathing training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effectiveness of receiving abdominal breathing training (Experimental): The patients receiving the intervention of abdominal breathing training were in the experimental group. The experimental group received the abdominal breathing training for a total of 8 weeks. During this period, they received the abdominal breathing training at the outpatient clinic (every day 30 minutes, can include every time during the day). When the subjects were at home, they received self-training using the abdominal breathing training video (once every day and 30 minutes every time). The control group without training.
  Interventions: Other: abdominal breathing training
- The effectiveness of not receiving abdominal breathing training (No Intervention): The control group who did not receive abdominal breathing training. The effectiveness assessment used the Beck anxiety inventory and physiological index (heart beats, breath and blood pressure), required to be completed by the control group.

INTERVENTIONS:
Other: abdominal breathing training — The abdominal breathing training at the outpatient clinic (every day 30 minutes, can include every time during the day). When the subjects were at home, they received self-training using the abdominal breathing training video (once every day and 30 minutes every time).
  Arms: The effectiveness of receiving abdominal breathing training

SUMMARY:
The research purpose is to investigate the effectiveness of abdominal breathing training on reducing anxiety. This study is an experimental research design. Using a randomized controlled trial approach. The patients receiving the intervention of abdominal breathing training were in the experimental group, while those who did not receive it were in the control group.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effectiveness of the abdominal breathing training on reducing anxiety. Using an experimental randomized controlled trial approach. The experimental group receiving abdominal breathing training, and control group without training. The effectiveness assessment used the Beck anxiety inventory, required to be completed by both the experimental group and control group. This study performed the pre-and-post assessments. This study performed the pre-test before the implementation of abdominal breathing training, and performed the post-test at Week 4 and Week 8 the end of abdominal breathing training. During this period, they received the abdominal breathing training at the outpatient clinic (every day 30 minutes, can include every time during the day). When the subjects were at home, they received self-training using the abdominal breathing training video (once every day and 30 minutes every time).

ELIGIBILITY:
Inclusion Criteria:

1. Who are over 20 years old.
2. The score of Beck anxiety inventory at lease of 8.
3. Agree to participate in the study and have filled out a written consent form.

Exclusion Criteria:

1. Inpatients.
2. COPD patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Beck anxiety inventory | pretest
  The total items of Beck anxiety inventory are 21. The score of each item is from 0-3. The score 0-7 is the least mild anxiety, 8-15 is the mild anxiety, 16-25 is the moderate anxiety, and 26-63 is the severe anxiety
Beck anxiety inventory | post-test at Week 4
  The total items of Beck anxiety inventory are 21. The score of each item is from 0-3. The score 0-7 is the least mild anxiety, 8-15 is the mild anxiety, 16-25 is the moderate anxiety, and 26-63 is the severe anxiety
Beck anxiety inventory | post-test at Week 8
  The total items of Beck anxiety inventory are 21. The score of each item is from 0-3. The score 0-7 is the least mild anxiety, 8-15 is the mild anxiety, 16-25 is the moderate anxiety, and 26-63 is the severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Xuan-Yi Huang, DNSc, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Xuan-Yi Huang, Taipei, Peitou, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cahalin LP, Braga M, Matsuo Y, Hernandez ED. Efficacy of diaphragmatic breathing in persons with chronic obstructive pulmonary disease: a review of the literature. J Cardiopulm Rehabil. 2002 Jan-Feb;22(1):7-21. doi: 10.1097/00008483-200201000-00002. PMID 11839992
- [Result] Chen YF, Huang XY, Chien CH, Cheng JF. The Effectiveness of Diaphragmatic Breathing Relaxation Training for Reducing Anxiety. Perspect Psychiatr Care. 2017 Oct;53(4):329-336. doi: 10.1111/ppc.12184. Epub 2016 Aug 23. PMID 27553981
- [Result] Gosselink RA, Wagenaar RC, Rijswijk H, Sargeant AJ, Decramer ML. Diaphragmatic breathing reduces efficiency of breathing in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1995 Apr;151(4):1136-42. doi: 10.1164/ajrccm.151.4.7697243.
- [Result] Hopper SI, Murray SL, Ferrara LR, Singleton JK. Effectiveness of diaphragmatic breathing for reducing physiological and psychological stress in adults: a quantitative systematic review. JBI Database System Rev Implement Rep. 2019 Sep;17(9):1855-1876. doi: 10.11124/JBISRIR-2017-003848. PMID 31436595
- See also: This article reviews the literature regarding the efficacy of DB in persons with chronic obstructive pulmonary disease (COPD), and reports on the beneficial and detrimental effects of DB in persons with COPD. — https://pubmed.ncbi.nlm.nih.gov/11839992/
- See also: The findings provide guidance for providing quality care that effectively reduces the anxiety level of care recipients in clinical and community settings. — https://pubmed.ncbi.nlm.nih.gov/27553981/
- See also: Tidal volume, respiratory frequency, and duty cycle did not change significantly during diaphragmatic breathing. Dyspnea sensation tended to increase during diaphragmatic breathing. — https://pubmed.ncbi.nlm.nih.gov/7697243/
- See also: The evidence suggests that diaphragmatic breathing may decrease stress as measured by physiologic biomarkers, as well psychological self-report tools. — https://pubmed.ncbi.nlm.nih.gov/31436595/